CLINICAL TRIAL: NCT02529982
Title: The Effect of Curcumin Supplementation on Anthropometric Indices, Insulin Resistance and Oxidative Stress in Patients With Type 2 Diabetes
Brief Title: Curcumin Supplementation and Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1370
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Non Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Active Comparator): 500 mg curcumin capsule
  Interventions: Dietary Supplement: Curcumin
- control (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin
  Arms: intervention
Dietary Supplement: Placebo
  Arms: control

SUMMARY:
Diabetes mellitus is the most common endocrine disorder, causes many complications such as micro- and macro-vascular diseases. Various kinds of antidiabetic drugs have been developed, but most of them have side effects. Recently, the use of natural plant products has gained more attention among scientists in order to prevent diabetic vascular complications. Curcumin is a natural yellow product derived from the turmeric rhizome which has shown to be non-toxic and exhibits various bio¬logical activities such as anti-oxidant, anti-inflammatory, anti-carcinogenic, and anti-diabetic effects. Curcumin is effective in reducing glycemic index and hyperlipidemia in rodent models and is relatively inexpensive and safe. Most of the studies conducted on animal model, and just a few of them are on human model. The present study was planned to evaluate the effects of curcumin supplementation The effect of curcumin supplementation on anthropometric indices, insulin resistance and oxidative stress in patients with type 2 diabetes

ELIGIBILITY:
insulin Inclusion Criteria:

* a) Tendency to participate b) Age range of 40-65 c) Suffering from diabetes type 2 ( between 1 to 10 yeares) d) BMI 18/5-30 e) Patients with diabetes who administer oral hypoglycemic agents and do not use

Exclusion Criteria:

* a) patients with liver diseases b) patients with kidney diseases c) patients with inflammatory diseases d) patients with liver diseases e) Administering herbal agents f) Administering multivitamins and minerals in past 3 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
fasting blood sugar | 10 weeks
Insulin | 10 week
HbA1c | 10 week
Homeostatic Model Assessment of Insulin Resistance | 10 week
Change in pancreatic B-cell function | 10 week

SECONDARY OUTCOMES:
total capacity antioxidant | 10 weeks
Malondialdehyde | 10 week
Body mass index | 10 week
Waist circumference | 10 week

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Iran